CLINICAL TRIAL: NCT06661746
Title: Multimodal Intravenous Analgesia Using Half-dose of Ketamine, Lidocaine and Magnesium Sulfate Provides Efficient Postoperative Analgesia for Patients Undergoing Major Abdominal Surgery: Randomized, Case-controlled Study
Brief Title: Efficient Postoperative Pain Management With Multimodal IV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Eman M Elafifi, Lecturer of Anesthesia, Pain & ICU, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rc 1-7-2024
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Analgesia, Epidural

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal Group (Active Comparator)
  Interventions: Drug: Multimodal IV analgesia
- Epidural Group (Active Comparator)
  Interventions: Drug: epidural analgesia

INTERVENTIONS:
Drug: Multimodal IV analgesia — Multimodal IV analgesia of lidocaine, ketamine and MS
  Arms: Multimodal Group
Drug: epidural analgesia — Opioid-based and epidural analgesia
  Arms: Epidural Group

SUMMARY:
Postoperative pain remains a prevalent concern despite ongoing improvements in surgical methods and pain management strategies. Opioids, while commonly prescribed, frequently lead to undesirable side effects. Epidural analgesia, though a viable option, carries its risks and complications. Recent research indicates that combining intravenous lidocaine and ketamine can significantly alleviate postoperative pain and decrease the reliance on opioids within the initial 24 hours following surgery. This approach offers a promising alternative with minimal additional adverse effects, suggesting a potential shift in pain management practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients were assigned for surgical intervention;
* Patients of ASA grade I-III;
* Patients were free of exclusion criteria;

Exclusion Criteria:

* Patients who are not in ASA grade I-III;
* Patients who had uncontrolled hypertension and/or diabetes mellitus;
* Patients who had uncompensated cardiac, renal, or hepatic diseases;
* Patients with coagulopathy, spinal deformity, allergy, or contraindication for the used drugs;
* Patients who refused to sign the informed consent were excluded from the study.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Proportion of patients reporting at least a 50% reduction in pain (measured by Numerical Rating Scale) in post-Operative follow up. | 3 months
  Value of Multimodal injection in Pain Reduction post operatively manifested by recurrence of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Banhā, El Qalyoubia, Egypt